CLINICAL TRIAL: NCT03291457
Title: A Prospective Non-Interventional Study to Evaluate the Use of Glucocorticoids in Combination With Tocilizumab in Daily Clinical Practice
Brief Title: A Study to Evaluate the Use of Glucocorticoids in Combination With Tocilizumab in Daily Clinical Practice
Acronym: COGNOS
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML39114
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (1):
- Glucocorticoids + Tocilizumab: Participants with RA who are receiving glucocorticoid treatment will be observed for up to 52 weeks after starting tocilizumab.
  Interventions: Drug: Tocilizumab; Drug: Glucocorticoid Agent

INTERVENTIONS:
Drug: Tocilizumab — For intravenous (IV) tocilizumab, the recommended dosage is 8 milligrams per kilogram (mg/kg) once every 4 weeks. For subcutaneous (SC) tocilizumab, the recommended dosage is 162 milligrams (mg) once weekly. However, because of the observational nature of the study, dosing and treatment duration is at the discretion of the physician in accordance with local clinical practice and local labeling.
  Other Names: RoActemra
Drug: Glucocorticoid Agent — Because of the observational nature of the study, the choice of glucocorticoid agent, as well as dosing and treatment duration, is at the discretion of the physician in accordance with local clinical practice and local labeling.

SUMMARY:
This prospective, multicenter, observational study will evaluate the use of concomitant glucocorticoid therapy in adults with rheumatoid arthritis (RA) being treated with tocilizumab in daily clinical practice. Participants will be observed for up to 52 weeks after starting treatment with tocilizumab. All visits and assessments will be performed as per routine clinical practice, with no study-specific visits or interventions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe RA, defined as DAS28 greater than or equal to 3.7
* Naive to tocilizumab, or received tocilizumab within 8 weeks prior to enrollment
* Physician has made decision to commence IV or SC tocilizumab in accordance with label and reimbursement criteria
* Treated with glucocorticoids for RA when starting tocilizumab treatment

Exclusion Criteria:

* Treatment with any investigational agent within 4 weeks or 5 half-lives before tocilizumab
* Continuous or regular treatment with oral corticosteroids for any indication other than RA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will follow participants with RA who are receiving glucocorticoids prior to start of tocilizumab in daily clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2017-03-30 (Actual); Primary Completion 2019-12-04 (Actual); Study Completion 2019-12-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Are Able to Discontinue Use of Glucocorticoid without Loss of Disease Control According to Disease Activity Score Based on 28 Joints (DAS28) | Week 52
Percentage of Participants Who Are Able to Reduce Use of Glucocorticoid by 50 Percent (%) or More without Loss of Disease Control According to DAS28 | Week 52
Percentage of Participants by Reason for Glucocorticoid Dose Modification | Baseline up to Week 52

SECONDARY OUTCOMES:
Glucocorticoid Dose | Baseline; Weeks 24 and 52
Percentage of Participants Who Are Able to Reduce Use of Glucocorticoid by 25%, 50%, 75%, or 100% | Weeks 24 and 52
Percentage of Participants in Need of Glucocorticoid Dose Increase by 25%, 50%, 75%, or 100% | Weeks 24 and 52
Time to First Glucocorticoid Dose Reduction | Baseline up to Week 52
Time to Glucocorticoid Discontinuation | Baseline up to Week 52
Percentage of Participants in Remission According to DAS28 with Glucocorticoid Dose Reduction | Baseline up to Week 52
Percentage of Participants in Remission According to DAS28 with Glucocorticoid Dose Reduction of At Least 25%, 50%, or 75% | Baseline up to Week 52
Percentage of Participants in Remission According to DAS28 Who Discontinued Glucocorticoids | Baseline up to Week 52
Percentage of Participants with Low Disease Activity (LDA) According to DAS28 with Glucocorticoid Dose Reduction | Baseline up to Week 52
Percentage of Participants with LDA According to DAS28 with Glucocorticoid Dose Reduction of At Least 25%, 50%, or 75% | Baseline up to Week 52
Percentage of Participants with LDA According to DAS28 Who Discontinued Glucocorticoids | Baseline up to Week 52
Glucocorticoid Dose among Participants in Remission According to DAS28 | Baseline up to Week 52
Glucocorticoid Dose among Participants with LDA According to DAS28 | Baseline up to Week 52
Correlation between DAS28 Score and Glucocorticoid Dose | Baseline up to Week 52
Percentage of Participants with Adverse Events | Baseline up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- Belgium (22):
  - ASZ Aalst, Aalst
  - Onze Lieve Vrouwziekenhuis Aalst, Aalst
  - Dr. Huppertz - Marx pgmbh, Amel
  - Private Practice Els Van Essche, Bonheiden
  - AZ Sint Jan, Bruges
  - CHU St Pierre (César de Paepe), Brussels
  - Hospital Erasme, Brussels
  - Rhumarc sciv sprl, Céroux-Mousty
  - UZ Antwerpen, Edegem
  - Rhumaconsult sciv sprl; Private Practice, Forchies-la-Marche
  - Reumacentrum Genk, Genk
  - Reumaclinic, Genk
  - AZ Sint Lucas (Sint Lucas), Ghent
  - GHdC Site Saint-Joseph, Gilly (Charleroi)
  - Heilig Hartziekenhuis vzw, Lier
  - CHC MontLégia, Liège
  - CHU de Liège; Rhumatologie, Liège
  - Private Practice; Reumatologie, Mechelen
  - AZ Damiaan, Ostend
  - AZ Alma vzw (Sijsele), Sijsele
  - AZ Turnhout Sint Jozef, Turnhout
  - AZ Sint Jozef Malle, Westmalle